CLINICAL TRIAL: NCT01925352
Title: Phase 2 Study of Adenovirus Hepatocyte Growth Factor for Treatment of Ischemic Heart Disease
Brief Title: Safety Study of Adenovirus Hepatocyte Growth Factor to Treat Ischemic Heart Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Academy Military Medical Science, China (Industry)
Responsible Party: Principal Investigator, zhijian yang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIHD
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Heart Disease
Keywords: ischemic heart disease; adenovirus; hepatocyte growth factor
MeSH Terms: conditions — Myocardial Ischemia; Adenoviridae Infections; Deafness, Autosomal Recessive 39

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-HGF (Experimental): 5×10(9)pfu adenovirus hepatocyte growth factor was delivered by transendocardial injection in patients with ischemic heart disease into five left ventricular sites once.
  Interventions: Drug: Ad-HGF

INTERVENTIONS:
Drug: Ad-HGF — 5×10(9)pfu adenovirus hepatocyte growth factor was delivered by transendocardial injection into five left ventricular sites.
  Other Names: adenovirs hepatocyte growth factor

SUMMARY:
To explore the safety and efficiency of adenovirus-hepatocyte growth factor(Ad-HGF) treatment in ischemic heart disease.

DETAILED DESCRIPTION:
1. Ischemic heart disease refers to a group of closely related syndromes by an imbalance between the myocardial oxygen demand and the blood supply.
2. Gene therapy offers an attractive alternative to current pharmacologic therapies and may be beneficial in refractory disease. Gene therapy with hepatocyte growth factor induces angiogenesis, decreases apoptosis and leads to protection in the ischemic heart. In this study, we mainly explore the safety and effects of adenovirus hepatocyte growth factor for the treatment of ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* person with ischemic heart disease;
* Male or female of 20 to 70 years old;
* No blood perfusion detected in some area of heart using Single-Photon Emission Computed Tomography(SPECT) or Magnetic Resonance Imaging(MRI)
* two or more than two coronary arteries lesions were detected using coronary artery angiography and at least one coronary artery are un-suitable for percutaneous coronary intervention (PCI) or Coronary artery bypass grafting (CABG)；Or patients refuse to perform PCI or CABG
* LVEF is ≤45%;
* Patients must sign approved informed consent.

Exclusion Criteria:

* Acute myocardial infarction occured within one week
* CABG performed within 6 months or PCI performed within 3 months
* Patients with systemic active infection
* Blood alanine aminotransferase (ALT)>135mmol/L or blood crea(Cr)>200umol/L or patients with chronic obstructive pulmonary disease (COPD)
* patients with obvious bleeding tendency and blood disease
* patients with malignant tumor or end-stage disease
* patient anticipated life expectancy is less than 12 months
* patient recently attended test drugs or other device research

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with death,new myocardial infarction or stroke | 6 months after treatment

SECONDARY OUTCOMES:
left ventricular ejection fraction (LVEF) | 6 months after treatment

OTHER OUTCOMES:
tumor markers of blood | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Yang, PhD., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China